CLINICAL TRIAL: NCT00190489
Title: Phase III Trial of Doxorubicin /Cyclophosphamide (AC), Docetaxel (D), and Alternating AC and D (AC-D) as Front-line Chemotherapy for Metastatic Breast Cancer: Japan Clinical Oncology Group Trial (JCOG9802)
Brief Title: A Trial of Doxorubicin/Cyclophosphamide (AC), Docetaxel (D), and Alternating AC and D for Metastatic Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Japan Clinical Oncology Group (Other)
Collaborators: Ministry of Health, Labour and Welfare, Japan (Other Government)
Responsible Party: Japan Clinical Oncology Group, Japan Clinical Oncology Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JCOG9802; C000000179
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-08

CONDITIONS: Breast Cancer; Neoplasm Metastasis
Keywords: metastatic breast cancer; drug therapy; doxorubicin; docetaxel
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: AC (ADM 40mg/m2+CPA 500mg/m2) q21 days x 6 cycles
Drug: Docetaxel 60mg/m2 every 21 days for 6 cycles
Drug: AC and Docetaxel 60mg/m2 alternately q21 days for 6 cycles

SUMMARY:
To investigate the clinical benefits of Docetaxel or alternating AC-Docetaxel in comparison with standard AC for metastatic breast cancer

DETAILED DESCRIPTION:
power to detect a 50% increase in median TTF at 0.025 one-sided alpha in AC vs. D and AC vs. AC-D.

Results: 441pts (146 in AC, 147 in D, 148 in AC-D) were randomized between 01/99 and 05/03. Major grade 3-4 toxicities were neutropenia (26/45/46% for AC/D/AC-D), febrile neutropenia (3/4/6%), nausea/vomiting (3/3/4%). There was no toxic death. One grade 4 diarrhea in AC-D and 1 secondary leukemia (APL) in D were reported. Response (CR/PR) rates were 30, 41, and 35% for AC, D, and AC-D respectively. Median TTF (AC, D, and AC-D) are 6.4, 6.4, and 6.7 months (p =.255 for AC vs. D, p =.275 for AC vs. AC-D), and median overall survival are 22.4, 25.7, and 25.0 months (p=.092 for AC vs. D, p=.076 for AC vs. AC-D). The same difference was shown by the adjusted Cox model.

Conclusions: No benefit was demonstrated in D and AC-D over AC in TTF, however, D and AC-D tended to be superior to AC in response rate and overall survival. Survival benefit of front-line docetaxel should be re-evaluated by further long follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Hormonal therapy-resistant MBC
2. ER (-), failure of hormonal therapy for MBC, or relapse within 6 months after adjuvant hormonal therapy
3. No anthracyclines for MBC and no prior taxanes
4. At least 6 months from the completion of adjuvant chemotherapy
5. Measurable or evaluable lesions
6. Age: 20 to 75 years
7. PS: 0-3
8. WBC >= 4,000 /mm3 or ANC >=1,000 /mm3, Platelet >= 100,000 /mm3, SGOT/SGPT <= 1.5 x ULN, T-Bil <= 1.5 mg/dL, Cr <= 1.5 mg/dL
9. normal ECG
10. Written informed consent

Exclusion Criteria:

1. pregnant
2. malignant pleural effusion, ascites, or pericardial effusion that requires emergent treatment
3. Active infection
4. other cancer present within the last 5 years
5. previous stem cell transplantation
6. brain metastasis that requires emergent treatment
7. relapse within 6 months after completion anthracycline or during anthracycline
8. more than 250mg/m2 of anthracyclines
9. hypersensitivity of drug
10. interstitial pneumonitis or pulmonary fibrosis
11. positive HBs
12. antipsychotic medication
13. doctor's judgement

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450
Dates: Start 1999-01; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
time to treatment failure

SECONDARY OUTCOMES:
overall survival
progression-free survival
response rate
adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Shigemitsu Takashima, MD, PhD, Study Chair — National Shikoku Cancer Center
Locations (1):
- National Cancer Center Hospital, Chuo-ku, Tsukiji, 5-1-1, Tokyo, Japan

REFERENCES:
- See also: Related Info — http://www.jcog.jp/